CLINICAL TRIAL: NCT07254819
Title: The Effect of Cotinus Coggygria Mouthwash on Halitosis and Oral Hygiene in Orthodontic Patients: a Randomized Clinical Trial
Brief Title: Cotinus Coggygria Mouthwash and Halitosis and Oral Hygiene in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Iosif Sifakakis, Associate Professor, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 680/03.02.2025
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Orthodontic Appliance Complication; Halitosis
Keywords: halitosis; Cotinus Coggygria; Orthodontic Appliance
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Intervention Model Description: This trial is designed as a prospective, randomized, placebo-controlled, double (investigator and patient) blinded study, with two parallel groups and an equal allocation ratio in all groups. In this study, the intervention consists of delivery of Cotinus Coggygria mouthwash or placebo mouthwash.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All patients will be allocated at a 1:1 ratio between group A (Cotinus Coggygria group) and group B (placebo group), for each sex separately using stratified randomization. Two random sequences of 15 letters (A or B) will be obtained from www.random.org (List Randomizer service), one for males and one for females. Those letters were written on paper and then sealed in opaque envelopes, sequentially numbered from M1 to M15 for males and from F1 to F15 for females respectively. All envelopes were sealed, numbered and stored in a drawer by a person not involved in the study. Every patient enrolled in the study will receive an envelope in a numerical order and their name was written on the envelope. Informed consent will be obtained from parents / legal guardians and written consent upon information and prior to the randomization or application of any procedure obtained from the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Experimental group Cotinus Coggygria mouthwash (Experimental): Experimental Group: patients, age 13-18, conventional brackets, Cotinus Coggygria mouthwash 15 patients, with conventional brackets
  Interventions: Dietary Supplement: Cotinus Coggygria mouthwash
- Placebo control arm: placebo mouthwash (Placebo Comparator): Control Group: patients, age 13-18, conventional brackets, Placebo mouthwash 15 patients, with conventional brackets
  Interventions: Dietary Supplement: Placebo mouthwash

INTERVENTIONS:
Dietary Supplement: Cotinus Coggygria mouthwash — All 30 patients will be randomly assigned to either the Cotinus Coggygria mouthwash group A (Natural Smoke Tree Hydrolina, Ina Essentials) (n = 15) or the placebo Mouthwash group B (from the same manufacturer) (n = 15). All patients will be asked to use the mouthwash twice a day for 14 days and to maintain their usual oral hygiene routine. The measurements will be done in the morning and at least three hours after brushing and without the use of the mouthwash by the participant on the day of the assessments.
  Arms: Experimental: Experimental group Cotinus Coggygria mouthwash
Dietary Supplement: Placebo mouthwash — All 30 patients will be randomly assigned to either the group A (Cotinus Coggygria mouthwash ) (n = 15) or the placebo Mouthwash group B (from the same manufacturer) (n = 15). All patients will be asked to use the mouthwash twice a day for 14 days and to maintain their usual oral hygiene routine. The measurements will be done in the morning and at least three hours after brushing and without the use of the mouthwash by the participant on the day of the assessments.
  Arms: Placebo control arm: placebo mouthwash

SUMMARY:
The aim of this trial was to investigate the effect of Cotinus Coggygria mouthwash on halitosis using as proxy the levels of the Volatile Sulfur Compounds (VSCs), and the effect on plaque and gingival indices in adolescents undergoing orthodontic treatment with fixed conventional labial appliances.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for the trial must comply with all of the following at randomization:

• Age between 13 and 18 years for the group with conventional orthodontic appliances.

This age group represents the majority of patients seeking orthodontic treatment and is homogeneous regarding occupational status (high-school and lyceum students in Greece). Younger patients might present with cooperation problems.

* Good general health.
* Orthodontic fixed labial appliances on the maxillary and mandibular arch, brackets at least on 20 teeth for more than 4 months before enrollment and estimated duration of the treatment more than 1 month, bands on the first molars, extraction cases patients could be enrolled at least two months after the last extraction.
* Total initial VSCs levels above the baseline level of 150ppb.

Exclusion Criteria:

Patients will be excluded for any of the following reasons:

* Active caries
* Periodontitis
* Dental fluorosis / dysplasia of the teeth
* Syndromes, mental disabilities and craniofacial deformities
* Smoking or use of other tobacco products
* Allergy to Cotinus Coggygria (Smoke tree)
* Antibiotics during the last 2 months
* Chlorhexidine or other mouthwash use in the previous 3 weeks
* Participation in other trials

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2025-12-03 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Hydrogen Sulfide (H2S) Levels | baseline
  Halitosis can be assessed using Gas chromatography that offers highly accurate qualitative and quantitative analysis of the individual VSCs, making it the preferred method for comprehensive diagnostic evaluation in both routine and complex cases. Halitosis is typically defined by a total VSCs concentration of ⩾150 ppb, a threshold supported across multiple clinical studies.
  The malodor results from the degradation of organic components in saliva, leading to the production of volatile sulfur compounds (VSCs), including hydrogen sulfide (H2S). H2S has been linked to increased gingival cell apoptosis and susceptibility to periodontitis.
Hydrogen Sulfide (H2S) Levels | 2 weeks
  Halitosis can be assessed using Gas chromatography that offers highly accurate qualitative and quantitative analysis of the individual VSCs, making it the preferred method for comprehensive diagnostic evaluation in both routine and complex cases. Halitosis is typically defined by a total VSCs concentration of ⩾150 ppb, a threshold supported across multiple clinical studies.
  The malodor results from the degradation of organic components in saliva, leading to the production of volatile sulfur compounds (VSCs), including hydrogen sulfide (H2S). H2S has been linked to increased gingival cell apoptosis and susceptibility to periodontitis.

SECONDARY OUTCOMES:
Modified plaque index (PI-M) | baseline
  The Silness and Löe index (Silness and Löe, 1964) does not take into account the pattern of plaque accumulation in orthodontic patients. To overcome this problem, Williams et al. (1991) divided the tooth into mesial, distal, gingival, and incisal regions in relation to the bracket and scored plaque in each region using the four codes of the original index (0 to 3). The values are summed to obtain a total score, which ranges from 0 to 12 for each tooth. This modified index is recommended for patients with fixed orthodontic appliances because it acknowledges the usual effects of orthodontic appliances on plaque distribution and has much greater categorical discrimination.
Modified plaque index (PI-M) | 2 weeks
  The Silness and Löe index (Silness and Löe, 1964) does not take into account the pattern of plaque accumulation in orthodontic patients. To overcome this problem, Williams et al. (1991) divided the tooth into mesial, distal, gingival, and incisal regions in relation to the bracket and scored plaque in each region using the four codes of the original index (0 to 3). The values are summed to obtain a total score, which ranges from 0 to 12 for each tooth. This modified index is recommended for patients with fixed orthodontic appliances because it acknowledges the usual effects of orthodontic appliances on plaque distribution and has much greater categorical discrimination.
Gingival Index (GI) | baseline
  The original Silness and Löe Plaque Index (1964) was not designed for orthodontic patients. The present study adopted a widely used modification of this index, in which the teeth are divided into incisal, distal, and mesial areas relative to the bracket, and plaque is graded in each area using values from 0 to 3.
Gingival Index (GI) | 2 weeks
  The original Silness and Löe Plaque Index (1964) was not designed for orthodontic patients. The present study adopted a widely used modification of this index, in which the teeth are divided into incisal, distal, and mesial areas relative to the bracket, and plaque is graded in each area using values from 0 to 3.
Dimethyl Sulfide [ (CH3)2S] Levels | baseline
  Halitosis can be assessed using Gas chromatography that offers highly accurate qualitative and quantitative analysis of the individual VSCs, making it the preferred method for comprehensive diagnostic evaluation in both routine and complex cases. Halitosis is typically defined by a total VSCs concentration of ⩾150 ppb, a threshold supported across multiple clinical studies. The malodor results from the degradation of organic components in saliva, leading to the production of volatile sulfur compounds (VSCs), including Dimethyl Sulfide [ (CH3)2S] Levels.
Dimethyl Sulfide [ (CH3)2S] Levels | 2 weeks
  Halitosis can be assessed using Gas chromatography that offers highly accurate qualitative and quantitative analysis of the individual VSCs, making it the preferred method for comprehensive diagnostic evaluation in both routine and complex cases. Halitosis is typically defined by a total VSCs concentration of ⩾150 ppb, a threshold supported across multiple clinical studies. The malodor results from the degradation of organic components in saliva, leading to the production of volatile sulfur compounds (VSCs), including Dimethyl Sulfide [ (CH3)2S] Levels.
Methyl-mercaptan (CH3SH) Levels | baseline
  Halitosis can be assessed using Gas chromatography that offers highly accurate qualitative and quantitative analysis of the individual VSCs, making it the preferred method for comprehensive diagnostic evaluation in both routine and complex cases. Halitosis is typically defined by a total VSCs concentration of ⩾150 ppb, a threshold supported across multiple clinical studies. The malodor results from the degradation of organic components in saliva, leading to the production of volatile sulfur compounds (VSCs), including Methyl-mercaptan (CH3SH) levels.
Methyl-mercaptan (CH3SH) Levels | 2 weeks
  Halitosis can be assessed using Gas chromatography that offers highly accurate qualitative and quantitative analysis of the individual VSCs, making it the preferred method for comprehensive diagnostic evaluation in both routine and complex cases. Halitosis is typically defined by a total VSCs concentration of ⩾150 ppb, a threshold supported across multiple clinical studies. The malodor results from the degradation of organic components in saliva, leading to the production of volatile sulfur compounds (VSCs), including Methyl-mercaptan (CH3SH) levels.

CONTACTS AND LOCATIONS:
Overall Officials: Iosif Sifakakis, Associate Professor, Study Director — National and Kapodistrian University of Athens, Greece
Locations (1):
- School of Dentistry, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No